CLINICAL TRIAL: NCT01808144
Title: A Long-Term Extension Study of Lesinurad in Combination With Febuxostat for Subjects With Gout Completing an Efficacy and Safety Study of Lesinurad and Febuxostat
Brief Title: Lesinurad and Febuxostat Combination Extension Study in Gout
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDEA594-307; 2012-004390-54 (EudraCT Number)
Record Dates: First submitted 2013-03-07; First posted 2013-03-11 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Gout
Keywords: Gout
MeSH Terms: conditions — Gout | interventions — lesinurad; Febuxostat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lesinurad 400 mg + febuxostat 80 mg (Experimental): Patients on lesinurad 400 mg had their dose changed to lesinurad 200 mg after implementation of protocol amendment 3, dated 07 October 2015.
  Interventions: Drug: lesinurad; Drug: febuxostat
- lesinurad 200 mg + febuxostat 80 mg (Experimental)
  Interventions: Drug: lesinurad; Drug: febuxostat

INTERVENTIONS:
Drug: lesinurad — Tablets, 400 mg once daily (QD)
  Arms: lesinurad 400 mg + febuxostat 80 mg
Drug: lesinurad — Tablets, 200 mg QD
  Arms: lesinurad 200 mg + febuxostat 80 mg
Drug: febuxostat — Tabletsm 80 mg QD

SUMMARY:
This study will assess the serum uric acid lowering effects and safety of lesinurad in combination with febuxostat over a long-term timeframe.

DETAILED DESCRIPTION:
This is a Phase 3 extension study to assess the long-term efficacy and safety of lesinurad in combination with febuxostat in subjects who completed the double-blind treatment period in Study RDEA594-304.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to understand the study procedures and the risks involved and is willing to provide written informed consent before the first study related activity.
* Subject completed the double-blind treatment period in Study RDEA594-304 and was actively receiving and tolerating study medication (lesinurad or placebo) and febuxostat 80 mg at the Month 12 visit.
* Subject is male or female; female subjects of childbearing potential must agree to use an effective non-hormonal method of birth control during the study and for at least 14 days after the last dose of study medication.

Exclusion Criteria:

* Subject has any medical or psychological condition, which in the opinion of the Investigator and/or the Medical Monitor, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements, or to complete the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2016-08-09 (Actual); Study Completion 2016-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nihar Bhakta, MD, Study Director — Ardea Biosciences, Inc.
Locations (68):
- United States (53):
  - Birmingham, Alabama
  - Tempe, Arizona
  - Glendale, California
  - Huntington Beach, California
  - Irvine, California
  - San Diego, California
  - Denver, Colorado
  - Englewood, Colorado
  - Boynton Beach, Florida
  - Naples, Florida
  - Pembroke Pines, Florida
  - Tampa, Florida
  - Winter Haven, Florida
  - Johns Creek, Georgia
  - Honolulu, Hawaii
  - Meridian, Idaho
  - Gurnee, Illinois
  - Springfield, Illinois
  - Elizabethtown, Kentucky
  - Frederick, Maryland
  - Ann Arbor, Michigan
  - Southfield, Michigan
  - Jackson, Mississippi
  - Olive Branch, Mississippi
  - Jefferson City, Missouri
  - St Louis, Missouri
  - New York, New York
  - Wilmington, North Carolina
  - Fargo, North Dakota
  - Columbus, Ohio
  - Middleburg Heights, Ohio
  - Wadsworth, Ohio
  - Oklahoma City, Oklahoma
  - Belle Vernon, Pennsylvania
  - Lansdale, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Sellersville, Pennsylvania
  - Columbia, South Carolina
  - Mt. Pleasant, South Carolina
  - Spartanburg, South Carolina
  - Memphis, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Victoria, Texas
  - Waco, Texas
  - Chesapeake, Virginia
  - Danville, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Morgantown, West Virginia
- Australia (3):
  - Camperdown, New South Wales
  - Woodville South, South Australia
  - Hobart, Tasmania
- Canada (2):
  - Mississauga, Ontario
  - Toronto, Ontario
- New Zealand (2):
  - Grafton, Auckland
  - Tauranga
- Poland (7):
  - Poznan, Greater Poland Voivodeship
  - Kutno, Iodzkie
  - Krakow, Lesser Poland Voivodeship
  - Bialystok, Podlaskie Voivodeship
  - Katowice, Silesian Voivodeship
  - Elblag, Warmian-Masurian Voivodeship
  - Gmina Końskie, Świętokrzyskie Voivodeship
- Fribourg, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects entered this extension Study RDEA594-307 while the core Study RDEA594-304 was ongoing and the database was not yet locked. To maintain the blind of the core study for subjects entering the extension, the lesinurad dose for all subjects in this extension study was blinded to the Sponsor until database lock of Study RDEA594-304.
Pre-assignment Details: Subjects randomized to lesinurad (RDEA594) 200 mg or 400 mg + febuxostat (FBX) 80 mg in Study RDEA594-304 continued to receive the same dose in this study. Subjects randomized to placebo + febuxostat 80 mg in Study RDEA594-304 were randomized in a double-blind, 1:1 fashion to either lesinurad 200 mg or 400 mg + febuxostat 80 mg.
Period: Overall Study
Arm/Group | Lesinurad 200 mg + Febuxostat 80 mg | Lesinurad 400 mg + Febuxostat 80 mg
Started | 97 | 99
Completed | 57 | 51
Not Completed | 40 | 48
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 16 | 23
Not completed — Lost to Follow-up | 6 | 3
Not completed — Protocol Violation | 6 | 6
Not completed — Gout flare | 0 | 1
Not completed — Adverse Event | 11 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lesinurad 400 mg + Febuxostat 80 mg | Lesinurad 200 mg + Febuxostat 80 mg | Total
Number analyzed (Participants) | 99 | 97 | 196
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.1 (10.58) | 52.9 (10.24) | 52.5 (10.41)
Age, Customized [Number; unit: Participants]
  < 65 years | 88 | 87 | 175
  >=65 years | 11 | 10 | 21
Sex/Gender, Customized [Number; unit: Participant]
  Male | 7 | 1 | 8
  Female | 92 | 96 | 188
Region of Enrollment [Number; unit: Participants]
  United States | 72 | 72 | 144
  Canada | 2 | 6 | 8
  Poland | 12 | 13 | 25
  Switzerland | 1 | 0 | 1
  Australia | 5 | 3 | 8
  New Zealand | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an sUA Level That is < 5.0 mg/dL
Description: Percentage of participants in Study 307 With sUA < 5.0 mg/dL from the Core Studies 304 and Extension Study 307 - Observed Cases
Time Frame: Up to approximately 2.5 years (at Extension Month 12)
Population: Number of Participants Analyzed for this Outcome Measure reflects the number of participants who completed Extension Month 12.
Measure: Number; unit: Percentage of participants
Arm/Group | Lesinurad 400 mg + Febuxostat 80 mg | Lesinurad 200 mg + Febuxostat 80 mg
Number analyzed (Participants) | 80 | 72
Percentage of participants | 82.5 | 77.8

2. Secondary Outcome: Percentage of Participants (With at Least One Target Tophus at Baseline) Who Experience Complete Resolution of at Least One Target Tophus
Description: Percentage of participants (With at Least One Target Tophus at Baseline) Who Experience Complete Resolution of at Least One Target Tophus During the Core and Extension Studies at Extension Month 12 (Observed Cases)
Time Frame: Up to approximatley 2.5 years (at Extension Month 12)
Population: ITT Population Number of Participants Analyzed for this Outcome Measure reflects the number of participants who completed through Month 12.
Measure: Number; unit: Percentage of participants
Arm/Group | Lesinurad 400 mg + Febuxostat 80 mg | Lesinurad 200 mg + Febuxostat 80 mg
Number analyzed (Participants) | 77 | 70
Percentage of participants | 61.0 | 54.3

ADVERSE EVENTS:
Time Frame: Up to approximately 2.5 years (at Extension Month 12)
Arm/Group | Lesinurad 200 mg + Febuxostat 80 mg | Lesinurad 400 mg + Febuxostat 80 mg
All-Cause Mortality (participants affected / at risk) | 1/97 | 0/99
Serious Adverse Events (participants affected / at risk) | 16/97 | 19/99
Other Adverse Events (participants affected / at risk) | 61/97 | 70/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lesinurad 200 mg + Febuxostat 80 mg (N=97) | Lesinurad 400 mg + Febuxostat 80 mg (N=99)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Joint destruction (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Stag horn calculus (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than .05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lesinurad 200 mg + Febuxostat 80 mg (N=97) | Lesinurad 400 mg + Febuxostat 80 mg (N=99)
Blood creatinine increased (Investigations) | 11 (14) | 13 (15)
Nasopharyngitis (Infections and infestations) | 6 (6) | 14 (20)
Hypertension (Vascular disorders) | 6 (6) | 10 (10)
Bronchitis (Infections and infestations) | 11 (12) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 8 (10) | 6 (9)
Sinusitis (Infections and infestations) | 8 (8) | 5 (5)
Headache (Nervous system disorders) | 5 (6) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (10) | 5 (5)
Urinary tract infection (Infections and infestations) | 6 (11) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 6 (11)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4)
Toothache (Gastrointestinal disorders) | 4 (4) | 5 (5)
Creatinine renal clearance decreased (Investigations) | 5 (6) | 3 (3)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 6 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 4 (6)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 6 (7)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 6 (6)
Muscle strain (Injury, poisoning and procedural complications) | 6 (7) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Cellulitis (Infections and infestations) | 3 (3) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 5 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
C-reactive protein increased (Investigations) | 2 (3) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 4 (4)
Insomnia (Psychiatric disorders) | 4 (4) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Liver function test abnormal (Investigations) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 3 (5)
Tooth abscess (Infections and infestations) | 1 (1) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall submit a copy of the Publication to Sponsor for review at least 45 days prior to its proposed submission. Sponsor reserves the right to delay any such publication for an additional period of 60 days. Upon Sponsor's request, PI agrees to delete from the proposed publication any Confidential Information. PI agrees not to release any publication without the prior written permission of Sponsor.